CLINICAL TRIAL: NCT01258829
Title: British Randomised Controlled Trial of AV and VV Optimisation (BRAVO): Randomised Clinical Trial of the Effects of Non-invasive Haemodynamic Optimisation of Cardiac Resynchronisation Devices on Exercise Capacity
Brief Title: British Randomised Controlled Trial of Atrioventricular (AV) and Interventricular (VV) Optimisation (BRAVO)
Acronym: BRAVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10/H0803/86
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure
Keywords: Heart Failure Cardiac Resynchronisation Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-invasive haemodynamic optimisation (Experimental): Optimization of pressure production by the heart, as measured by systolic blood pressure in the systemic circulation
  Interventions: Other: Non-invasive haemodynamic optimisation
- ECHO optimisation (Active Comparator): Optimization of AV/VV delay using the guideline recommendations
  Interventions: Other: ECHO optimisation

INTERVENTIONS:
Other: Non-invasive haemodynamic optimisation — Comparing the method of non-invasive haemodynamic
  Arms: Non-invasive haemodynamic optimisation
Other: ECHO optimisation — Standard ECHO optimisation method
  Arms: ECHO optimisation

SUMMARY:
Many patients who have cardiac resynchronisation therapy (a type of pacemaker) implanted for heart failure do not have the settings of their device optimised. The most widely available method for optimisation uses flow measured using cardiac ultrasound (echocardiography) to determine the optimal settings. However, this is not frequently performed because it is time consuming and requires two skilled operators. In this study the investigators will test a new non-invasive method for optimisation, which utilises pressure measurements (non-invasive blood pressure measured from the finger).

Is optimising AV and VV delay using non-invasive haemodynamics at least equivalent, in terms of exercise capacity, to conventional echo optimisation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure due to systolic dysfunction
* Biventricular pacemaker implanted
* Give written informed consent

Exclusion Criteria:

* Lung disease or any condition that would preclude them from walking on a treadmill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2010-12; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Is optimising AV and VV delay using non-invasive haemodynamics at least equivalent, in terms of exercise capacity, to conventional echo optimisation | 6 months following the last follow-up of the last patient

SECONDARY OUTCOMES:
To determine whether pressure optimisation is at least equivalent to echo optimisation of flow: in terms resulting size of the heart in terms of quality of life scores in terms of blood marker of heart failure severity | 6 months following the last follow-up of the last patient

CONTACTS AND LOCATIONS:
Overall Officials: Dr Darrel Francis, Principal Investigator — Imperial College London
Locations (1):
- ICCH, Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Whinnett ZI, Sohaib SMA, Mason M, Duncan E, Tanner M, Lefroy D, Al-Obaidi M, Ellery S, Leyva-Leon F, Betts T, Dayer M, Foley P, Swinburn J, Thomas M, Khiani R, Wong T, Yousef Z, Rogers D, Kalra PR, Dhileepan V, March K, Howard J, Kyriacou A, Mayet J, Kanagaratnam P, Frenneaux M, Hughes AD, Francis DP. Multicenter Randomized Controlled Crossover Trial Comparing Hemodynamic Optimization Against Echocardiographic Optimization of AV and VV Delay of Cardiac Resynchronization Therapy: The BRAVO Trial. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 1):1407-1416. doi: 10.1016/j.jcmg.2018.02.014. Epub 2018 May 16. PMID 29778861
- [Derived] Jones S, Lumens J, Sohaib SMA, Finegold JA, Kanagaratnam P, Tanner M, Duncan E, Moore P, Leyva F, Frenneaux M, Mason M, Hughes AD, Francis DP, Whinnett ZI; BRAVO Investigators. Cardiac resynchronization therapy: mechanisms of action and scope for further improvement in cardiac function. Europace. 2017 Jul 1;19(7):1178-1186. doi: 10.1093/europace/euw136. PMID 27411361
- [Derived] Whinnett ZI, Sohaib SM, Jones S, Kyriacou A, March K, Coady E, Mayet J, Hughes AD, Frenneaux M, Francis DP; BRAVO Investigators. British randomised controlled trial of AV and VV optimization ("BRAVO") study: rationale, design, and endpoints. BMC Cardiovasc Disord. 2014 Apr 3;14:42. doi: 10.1186/1471-2261-14-42. PMID 24693953
- [Derived] Jones S, Shun-Shin MJ, Cole GD, Sau A, March K, Williams S, Kyriacou A, Hughes AD, Mayet J, Frenneaux M, Manisty CH, Whinnett ZI, Francis DP. Applicability of the iterative technique for cardiac resynchronization therapy optimization: full-disclosure, 50-sequential-patient dataset of transmitral Doppler traces, with implications for future research design and guidelines. Europace. 2014 Apr;16(4):541-50. doi: 10.1093/europace/eut257. Epub 2013 Sep 25. PMID 24068445